CLINICAL TRIAL: NCT06688929
Title: Psychosocial and Functional Interactions in the Characterization of Axial Spondyloarthritis
Brief Title: Psychosocial and Functional Factors in AxSpA
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Other Study IDs: 07
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Spondyloarthropathies; Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Axial Spondyloarthritis Patients: A cohort of adult patients diagnosed with axial spondyloarthritis (AxSpA) according to the Assessment of SpondyloArthritis International Society (ASAS) criteria. These patients will be evaluated to analyze the impact of psychosocial factors on disease progression, functionality, and quality of life.

SUMMARY:
This observational, cross-sectional study aims to characterize patients with axial spondyloarthritis (AxSpA) from a biopsychosocial perspective. The study examines the relationships between psychosocial factors (such as pain catastrophizing, kinesiophobia, and fear-avoidance beliefs) and clinical indicators of disease progression, including functional limitations and disease activity. The primary objective is to identify psychosocial predictors of functionality and disease activity in AxSpA patients, which may guide more personalized therapeutic interventions. Findings could provide insights into the combined effects of physical and psychological aspects on disease management, promoting a holistic approach to AxSpA care.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) diagnosed with axial spondyloarthritis (AxSpA) based on the Assessment of SpondyloArthritis International Society (ASAS) criteria.
* Experiencing symptoms of axial or peripheral involvement.
* A minimum score of 3/10 on the Numeric Pain Rating Scale (NPRS) during the initial assessment.

Exclusion Criteria:

* Individuals with other rheumatic or musculoskeletal conditions affecting the spine or joints (e.g., rheumatoid arthritis or osteoarthritis).
* History of spinal surgery or joint replacement surgery.
* Receipt of corticosteroid injections or other pharmacological treatments targeting inflammation within six weeks prior to data collection.
* Any ongoing medico-legal conflicts that could interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with axial spondyloarthritis who meet the inclusion criteria and are recruited from healthcare facilities specializing in the treatment of musculoskeletal conditions.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline (single assessment at the start of the study)
  This primary outcome measure will assess disease activity in patients with axial spondyloarthritis using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The BASDAI is a validated, self-reported measure that evaluates symptoms such as fatigue, spinal pain, joint pain, and morning stiffness on a scale from 0 to 10, where higher scores indicate higher disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline (single assessment at the start of the study)
  A self-reported index measuring functional limitations in ankylosing spondylitis patients. It evaluates the ability to perform daily activities, with scores ranging from 0 to 10, where higher scores indicate greater functional impairment.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Baseline
  An index measuring spinal mobility in ankylosing spondylitis, using measurements of lateral lumbar flexion, tragus-to-wall distance, cervical rotation, lumbar flexion (modified Schober test), and intermalleolar distance. Each component is scored on a continuous scale from 0 to 10.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  A numeric rating scale for pain, where patients rate their pain intensity on a scale from 0 to 10, with 0 meaning "no pain" and 10 "the worst pain imaginable."
Range of Motion (ROM) | Baseline
  Cervical range of motion will be measured using a goniometer for flexion/extension, lateral flexion, and rotation movements. Lumbar flexion will be assessed using the modified Schober test.
Pressure Pain Threshold (PPT) | Baseline
  Pressure pain threshold will be assessed at specific points, such as the upper trapezius, lumbar erector spinae at L3-L4, and epicondyle muscles, using a mechanical pressure algometer.
Cervical Joint Position Sense Error (JPSE) | Baseline
  Assesses cervical proprioceptive acuity by measuring the error in repositioning the head to a neutral posture.
Lumbar Repositioning Error (LRE) | Baseline
  Assesses lumbar proprioception by measuring the error in repositioning after flexing the lumbar spine to a specific angle.

OTHER OUTCOMES:
Pain Catastrophizing Scale (PCS) | Baseline
  A self-reported scale that measures catastrophic thinking related to pain, including thoughts and feelings associated with pain experiences. It consists of 13 items rated on a Likert scale from 0 to 4, with higher scores indicating greater catastrophizing.
Tampa Scale for Kinesiophobia (TSK-11) | Baseline
  A scale that measures fear of movement and re-injury, consisting of 11 items rated on a scale from 1 to 4, with higher scores indicating greater fear of movement.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Baseline
  A questionnaire that assesses fear-avoidance beliefs related to physical activity and work in individuals with musculoskeletal pain. It includes two subscales: one for physical activity (FABQ-PA) and another for work-related fear-avoidance (FABQ-W), with items rated on a scale from 0 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Badajoz, Spain